CLINICAL TRIAL: NCT02693041
Title: Pregnancy Complications - A Probiotic Interventional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bo Jacobsson, Clinical professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dnr. 929-11
Record Dates: First submitted 2015-10-12; First posted 2016-02-26 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Preeclampsia; Preterm Birth
Keywords: Probiotics; inflammation; immunological response; preterm birth; preeclampsia
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Inflammation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PROBIOTIC in low-risk women (Active Comparator): In low-risk women, probiotic group will be treated with the Active ingredient containing Lactobacillus rhamnosus (LGG) (> 10x8 CFU) during all pregnancy until delivery. Capsules contain maltodextrin, LGG and vegetal magnesium stearate.
  Interventions: Drug: probiotic
- PLACEBO in low-risk women (Placebo Comparator): In low-risk women, placebo group will be treated with the placebo ingredient during all pregnancy until delivery. The capsules of the placebo Group have similar content but lack the probiotic lactic acid bacteria which has been replaced by maltodextrin to make the mg amount equal.
  Interventions: Drug: placebo
- PROBIOTIC in women with a prior PTB (Active Comparator): In women with a prior preterm birth (PTB), probiotic Group will be treated with the Active ingredient containing Lactobacillus rhamnosus (LGG) (> 10x8 CFU) during all pregnancy until delivery. Capsules contain maltodextrin, LGG and vegetal magnesium stearate.
  Interventions: Drug: probiotic
- PLACEBO in women with a prior PTB (Placebo Comparator): In women with a prior preterm birth (PTB), placebo group will be treated with the placebo ingredient during all pregnancy until delivery. The capsules of the placebo Group have similar content but lack the probiotic lactic acid bacteria which has been replaced by maltodextrin to make the mg amount equal.
  Interventions: Drug: placebo
- PROBIOTIC in women with a prior PE (Active Comparator): In women with a prior preeclampsia (PE), probiotic Group will be treated with the Active ingredient containing Lactobacillus rhamnosus (LGG) (> 10x8 CFU) during all pregnancy until delivery. Capsules contain maltodextrin, LGG and vegetal magnesium stearate.
  Interventions: Drug: probiotic
- PLACEBO in women with a prior PE (Placebo Comparator): In women with a prior preeclampsia (PE), placebo Group will be treated with the placebo ingredient during all pregnancy until delivery. The capsules of the placebo Group have similar content but lack the probiotic lactic acid bacteria which has been replaced by maltodextrin to make the mg amount equal.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: probiotic — Low-risk women, women with prior preeclampsia and women with a prior preterm birth will be randomized to be treated with LGG during pregnancy. Effect on maternal and perinatal outcome as well as the effect of treatment on immunological and inflammatory biomarkers will be evaluated.
  Other Names: Lactobacillus rhamnosus; LGG
  Arms: PROBIOTIC in low-risk women; PROBIOTIC in women with a prior PE; PROBIOTIC in women with a prior PTB
Drug: placebo — Low-risk women, women with prior preeclampsia and women with a prior preterm birth will be randomized to be treated with placebo during pregnancy. Effect on maternal and perinatal outcome as well as the effect of treatment on immunological and inflammatory biomarkers will be evaluated.
  Arms: PLACEBO in low-risk women; PLACEBO in women with a prior PE; PLACEBO in women with a prior PTB

SUMMARY:
Investigators hypothesize that

a) probiotics decrease the overall inflammatory state in the pregnant woman, especially in women with high risk pregnancies.

DETAILED DESCRIPTION:
The main of the Project is to determine if dietary supplementation intake of probiotics are associated with a decreased inflammatory response in pregnant women, especially those with a history of previous preterm birth or preeclampsia, in a randomized clinical trial. Investigators also want to further investigate the relationship between intake of probiotics and the degree of inflammation in different compartments during pregnancy to see how the probiotic components affect the inflammatory state in the women.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age > or = 18 y
* Singleton pregnancy
* Nulli or multiparous without maternal intercurrent diseases or pregnant women with a history of spontaneous preterm delivery or pregnant women with a history of preeclampsia.

Exclusion Criteria

* Multiple pregnancy
* Gestational age > 17+6 weeks at first visit
* Chronic intermittent diseases (e.g. diabetes mellitus, systemic lupus erythematosus, rheumatoid arthritis, Chron disease, ulcerative colitis)
* Uterus malformations
* Immunomodulatory medication
* Hormonal treatment (e.g. crinone, progesterone)
* Subject disagrees to stop intake of other products containing probiotics during study time.
* Subject is unable to provide written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Inflammatory modulation of Lactobacillus Rhamnosus in low risk mothers. | at recruitment, week 25, week 35 of gestation
  Intake of LGG Rhamnosus throughout the pregnancy and its effect on levels of subpopulations of lymphocytes in peripheral blood (T/B/NK-celler), and cytokine production (TNF alfa, IL10, IL12) after stimulation with E. Coli, L. paracasei and P. aerugnousa, measuring change from baseline to 25 and 35 weeks gestation.
Inflammatory modulation of Lactobacillus Rhamnosus in mothers with previous preterm birth. | at recruitment, week 25, week 35 of gestation
  Intake of LGG Rhamnosus throughout the pregnancy and its effect on levels of subpopulations of lymphocytes in peripheral blood (T/B/NK-celler), and cytokine production (TNF alfa, IL10, IL12) after stimulation with E. Coli, L. paracasei and P. aerugnousa, measuring change from baseline to 25 and 35 weeks gestation.
Inflammatory modulation of Lactobacillus Rhamnosus in mothers with previous preeclampsia. | at recruitment, week 25, week 35 of gestation
  Intake of LGG Rhamnosus throughout the pregnancy and its effect on levels of subpopulations of lymphocytes in peripheral blood (T/B/NK-celler), and cytokine production (TNF alfa, IL10, IL12) after stimulation with E. Coli, L. paracasei and P. aerugnousa, measuring change from baseline to 25 and 35 weeks gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Jacobsson, Professor, Principal Investigator — Göteborg University
Locations (1):
- Bo Jacobsson, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aagaard K, Ma J, Antony KM, Ganu R, Petrosino J, Versalovic J. The placenta harbors a unique microbiome. Sci Transl Med. 2014 May 21;6(237):237ra65. doi: 10.1126/scitranslmed.3008599. PMID 24848255
- [Result] Cobo T, Kacerovsky M, Palacio M, Hornychova H, Hougaard DM, Skogstrand K, Jacobsson B. Intra-amniotic inflammatory response in subgroups of women with preterm prelabor rupture of the membranes. PLoS One. 2012;7(8):e43677. doi: 10.1371/journal.pone.0043677. Epub 2012 Aug 20. PMID 22916296
- [Result] Goncalves LF, Chaiworapongsa T, Romero R. Intrauterine infection and prematurity. Ment Retard Dev Disabil Res Rev. 2002;8(1):3-13. doi: 10.1002/mrdd.10008. PMID 11921380
- [Result] Jimenez E, Fernandez L, Marin ML, Martin R, Odriozola JM, Nueno-Palop C, Narbad A, Olivares M, Xaus J, Rodriguez JM. Isolation of commensal bacteria from umbilical cord blood of healthy neonates born by cesarean section. Curr Microbiol. 2005 Oct;51(4):270-4. doi: 10.1007/s00284-005-0020-3. Epub 2005 Sep 20. PMID 16187156
- [Result] Jimenez E, Marin ML, Martin R, Odriozola JM, Olivares M, Xaus J, Fernandez L, Rodriguez JM. Is meconium from healthy newborns actually sterile? Res Microbiol. 2008 Apr;159(3):187-93. doi: 10.1016/j.resmic.2007.12.007. Epub 2008 Jan 11. PMID 18281199
- [Result] Myhre R, Brantsaeter AL, Myking S, Gjessing HK, Sengpiel V, Meltzer HM, Haugen M, Jacobsson B. Intake of probiotic food and risk of spontaneous preterm delivery. Am J Clin Nutr. 2011 Jan;93(1):151-7. doi: 10.3945/ajcn.110.004085. Epub 2010 Oct 27. PMID 20980489
- [Result] Brantsaeter AL, Myhre R, Haugen M, Myking S, Sengpiel V, Magnus P, Jacobsson B, Meltzer HM. Intake of probiotic food and risk of preeclampsia in primiparous women: the Norwegian Mother and Child Cohort Study. Am J Epidemiol. 2011 Oct 1;174(7):807-15. doi: 10.1093/aje/kwr168. Epub 2011 Aug 5. PMID 21821542
- [Result] Bertelsen RJ, Brantsaeter AL, Magnus MC, Haugen M, Myhre R, Jacobsson B, Longnecker MP, Meltzer HM, London SJ. Probiotic milk consumption in pregnancy and infancy and subsequent childhood allergic diseases. J Allergy Clin Immunol. 2014 Jan;133(1):165-71.e1-8. doi: 10.1016/j.jaci.2013.07.032. Epub 2013 Sep 10. PMID 24034345
- [Result] Yeganegi M, Watson CS, Martins A, Kim SO, Reid G, Challis JR, Bocking AD. Effect of Lactobacillus rhamnosus GR-1 supernatant and fetal sex on lipopolysaccharide-induced cytokine and prostaglandin-regulating enzymes in human placental trophoblast cells: implications for treatment of bacterial vaginosis and prevention of preterm labor. Am J Obstet Gynecol. 2009 May;200(5):532.e1-8. doi: 10.1016/j.ajog.2008.12.032. Epub 2009 Mar 14. PMID 19285652
- [Result] Yeganegi M, Leung CG, Martins A, Kim SO, Reid G, Challis JR, Bocking AD. Lactobacillus rhamnosus GR-1 stimulates colony-stimulating factor 3 (granulocyte) (CSF3) output in placental trophoblast cells in a fetal sex-dependent manner. Biol Reprod. 2011 Jan;84(1):18-25. doi: 10.1095/biolreprod.110.085167. Epub 2010 Sep 1. PMID 20811016

DOCUMENTS (1):
  • Informed Consent Form (2011-11-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT02693041/ICF_000.pdf